CLINICAL TRIAL: NCT01772797
Title: A Phase Ib, Open-label, Dose Escalation Study of LDK378 and AUY922 in Patients With ALK-rearranged Non-small Cell Lung Cancer
Brief Title: Phase Ib Study of LDK378 and AUY922 in ALK-rearranged Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378X2102; 2012-004632-29 (EudraCT Number)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-09

CONDITIONS: Anaplastic Lymphoma Kinase (ALK); Non-small Cell Lung Cancer
Keywords: anaplastic lymphoma kinase, ALK-rearranged lung cancer, non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ceritinib; 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDK378 and AUY922 (Experimental)
  Interventions: Drug: LDK378; Drug: AUY922

INTERVENTIONS:
Drug: LDK378 — LDK378 is a capsule to be taken daily by mouth.
Drug: AUY922 — AUY922 is an intravenous infusion that will be administered by the investigative site to the patient on a weekly basis.

SUMMARY:
The primary purpose of the study is to estimate the maximum tolerated dose of the combination of LDK378 and AUY922. This study will assess the safety, tolerability, pharmacokinetics and preliminary evidence of anti-tumor activity of the combination of LDK378 and AUY922 in ALK-rearranged non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* locally advanced or metastatic NSCLC that has progressed during or following therapy with an ALK inhibitor
* tumor must carry an ALK rearrangement in 15% or more of tumor cells as measured by FISH
* disease that can be evaluated by RECIST v1.1 and measurable disease

Exclusion Criteria:

* central nervous system (CNS) metastases that are symptomatic or require increasing steroids or CNS-directed therapy to control CNS disease
* history of interstitial lung disease or interstitial pneumonitis, including clinically significant radiation pneumonitis
* clinically significant cardiac dysfunction
* inadequate end organ function as defined by specified laboratory values
* use of medications known to be strong inhibitors or inducters of CYP3A4/5 that cannot be discontinued at least 1 week prior to start of treatment
* use of medications that are mainly metabolized by CYP3A4/5 or CYP2C9 that cannot be discontinued at least 1 week prior to start of treatment
* clinically significant, uncontrolled impaired gastrointestinal function or GI disease
* prior treatment with a HSP90 inhibitor
* radiotherapy to lung within 4 weeks prior to the first dose of study treatment or patients who have not recovered from radiotherapy-related toxicities
* pregnant or nursing women
* history of pancreatitis or history of increased amylase or lipase that was due to pancreatic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence rate of Dose Limiting Toxicities (DLT) | up to day 28 after the patient's first dose
  cycle = within the first 28 days of patient's first dose

SECONDARY OUTCOMES:
Number of patients with adverse events | 30 months
  Characterize the safety and tolerability of LDK378 and AUY922 in patients
Changes in laboratory values | 30 months
  Characterize the safety and tolerability of LDK378 and AUY922 in patients
Assessments of electrocardiograms | 30 months
  Characterize the safety and tolerability of LDK378 and AUY922 in patients
Assessments of dose interruptions, reductions, and dose intensity | 30 months
  Characterize the safety and tolerability of LDK378 and AUY922 in patients
Plasma PK parameter of LDK378 and AUY922: Tmax | 30 months
  Characterize single and multiple dose PK of LDK378 and AUY922 in patients
Overall response rate (ORR) | 30 months
  Assess the anti-tumor activity of LDK378 and AUY922
Duration of Response (DoR) | 30 months
  Assess the anti-tumor activity of LDK378 and AUY922
Time to Response (TTR) | 30 months
  Assess the anti-tumor activity of LDK378 and AUY922
Progression free survival (PFS) | 30 months
  Assess the anti-tumor activity of LDK378 and AUY922 per RECIST 1.1
Number of patients with serious adverse events | 30 months
  Characterize the safety and tolerability of LDK378 and AUY922 in patients
Plasma PK parameter of LDK378 and AUY922: Cmax | 30 months
  Characterize single and multiple dose PK of LDK378 and AUY922 in patients
Plasma PK parameter of LDK378 and AUY922: AUClast | 30 months
  Characterize single and multiple dose PK of LDK378 and AUY922 in patients
Plasma PK parameter of LDK378 and AUY922: AUCtau | 30 months
  Characterize single and multiple dose PK of LDK378 and AUY922 in patients
Plasma PK parameter of LDK378 and AUY922: Cmin | 30 months
  Characterize single and multiple dose PK of LDK378 and AUY922 in patients
Plasma PK parameter of LDK378 and AUY922: Racc | 30 months
  Characterize single and multiple dose PK of LDK378 and AUY922 in patients

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- United States (4):
  - University of Colorado Dept. of Anschutz Cancer (3), Aurora, Colorado
  - Massachusetts General Hospital Mass General, Boston, Massachusetts
  - Fox Chase Cancer Center Fox Chase Cancer (2), Philadelphia, Pennsylvania
  - University of Utah / Huntsman Cancer Institute Huntsman, Salt Lake City, Utah
- Novartis Investigative Site, Melbourne, Victoria, Australia
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain

REFERENCES:
- See also: Results for CLDK378X2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=15547